CLINICAL TRIAL: NCT01311648
Title: A Multicenter Phase III Uncontrolled Open-label Trial to Evaluate Safety and Efficacy of BAY81-8973 in Children With Severe Hemophilia A Under Prophylaxis Therapy
Brief Title: BAY81-8973 Pediatric Safety and Efficacy Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13400; 2010-021781-29 (EudraCT Number)
Record Dates: First submitted 2011-02-18; First posted 2011-03-09 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Haemophilia A
Keywords: Recombinant factor VIII; Pediatric use
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTPs 0-12 years (Experimental): Previously treated patients (PTPs) aged below 12 years received BAY81-8973 25-50 IU/kg at least 2x/week for 6 months and at least 50 exposure days (EDs) in main study - Part A. Participants having reached at least 50 EDs in main study - Part A were offered participation in an open label extension study (optional). Participants who transitioned from main study - Part A to the extension study received BAY81-8973, 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part A and extension study).
  Interventions: Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973)
- PUPs/MTPs 0-<6 years (Experimental): Previously untreated patients (PUPs) or minimally treated patients (MTPs, patients who had no more than 3 exposure days (EDs) with any FVIII product) received BAY81-8973 15-50 IU/kg at least 1x/week for at least 50 EDs or until inhibitor development in main study - Part B. Participants having reached at least 50 EDs in main study - Part B were offered participation in an open label extension study and received BAY81-8973 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part B and extension study); participants who developed an inhibitor in main study - Part B were offered participation in open label extension study and received Immune Tolerance Induction (ITI) treatment with BAY81-8973 until successful eradication of the inhibitor, or until failure, for approximately 18 months.
  Interventions: Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) — Main study: 25-50 IU/kg at least 2x/week for 6 months and at least 50 EDs, IV infusion; Extension study: 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part A and extension study), IV infusion. Exposure day (ED): An ED is a unit of time (1 day) in which replacement treatment of Hemophilia is given to a patient.
  Arms: PTPs 0-12 years
Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) — Main study: 15-50 IU/kg at least 1x/week for at least 50 EDs or until inhibitor development, IV infusion; Extension study: For participants having reached at least 50 EDs in main study - Part B: 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part B and extension study), IV infusion. For participants who developed an inhibitor in main study - Part B: up to 200 IU/kg per day or 100 IU/kg twice a day at the discretion of the investigator and coordinating investigator until successful eradication of the inhibitor, or until failure, for up to18 months (treatment beyond 18 months required an agreement with the sponsor and coordinating investigator), IV infusion
  Arms: PUPs/MTPs 0-<6 years

SUMMARY:
The primary objective was to evaluate the safety and efficacy of the treatment with BAY81-8973 for prophylaxis and treatment of breakthrough bleeds in children with severe hemophilia A.

The secondary objectives were

* To assess the safety and efficacy of BAY81-8973 during surgeries.
* To assess incremental recovery of BAY81-8973.
* To assess pharmacokinetic (PK) parameters in a subset of children (Previously treated patients [PTPs] and previously untreated patients [PUPs] / minimally treated patients [MTPs] - participation in PK sampling was voluntary and required consent).

ELIGIBILITY:
Inclusion Criteria:

* Male
* PTPs (previously treated patients): aged <= 12 years
* PUPs (previously untreated patients) / MTPs (minimally treated patients): aged < 6 years
* Severe hemophilia A defined as < 1% FVIII concentration (FVIII:C)
* PTPs: >= 50 exposure days (EDs) with any FVIII concentrate, no current evidence of inhibitory antibody, and no history of FVIII inhibitor formation
* PUPs: no prior exposure to any FVIII product
* MTPs: having no more than 3 EDs with any FVIII product, no current evidence of inhibitory antibody and no history of FVIII inhibitor formation

Exclusion Criteria:

* With another bleeding disorder that is different from Hemophilia A
* With thrombocytopenia (platelet count < 100 000/mm^3)
* Creatinine > 2x upper limit of normal or Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) > 5x upper limit of normal
* Without a negative inhibitor testing at screening (except for PUPs)
* Receiving chemotherapy, immune modulatory drugs, has received another investigational FVIII product within the last month, or received another experimental drug within the last 3 months
* Requires any pre-medication to tolerate FVIII treatment
* Known hypersensitivity to active substance, mouse, or hamster protein

Ages: 0 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2011-06-09 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (42):
- United States (4):
  - New Orleans, Louisiana
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
- Bahía Blanca, Buenos Aires, Argentina
- Bulgaria (2):
  - Plovdiv
  - Varna
- Canada (3):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Toronto, Ontario
- Århus N, Denmark
- Hungary (3):
  - Budapest
  - Debrecen
  - Mohács
- Crumlin, Dublin, Ireland
- Ramat Gan, Israel
- Italy (5):
  - Bari, Apulia
  - Rome, Lazio
  - Milan, Lombardy
  - Catania, Sicily
  - Padua, Veneto
- Riga, Latvia
- Vilnius, Lithuania
- Mexico (3):
  - Guadalajara, Jalisco
  - San Juan del Río, Querétaro
  - Oaxaca City
- Oslo, Norway
- Poland (3):
  - Lodz
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Timișoara
- Russia (3):
  - Kazan'
  - Kirov
  - Volgograd
- Spain (6):
  - Esplugues de Llobregat, Barcelona
  - A Coruña
  - Alicante
  - Cáceres
  - Madrid
  - Valencia

REFERENCES:
- [Result] Oldenburg J, Windyga J, Hampton K, Lalezari S, Tseneklidou-Stoeter D, Beckmann H, Maas Enriquez M. Safety and efficacy of BAY 81-8973 for surgery in previously treated patients with haemophilia A: results of the LEOPOLD clinical trial programme. Haemophilia. 2016 May;22(3):349-53. doi: 10.1111/hae.12839. Epub 2016 Mar 1. PMID 26931631
- [Result] Ljung R, Kenet G, Mancuso ME, Kaleva V, Rusen L, Tseneklidou-Stoeter D, Michaels LA, Shah A, Hong W, Maas Enriquez M; investigators of the LEOPOLD Kids Trial. BAY 81-8973 safety and efficacy for prophylaxis and treatment of bleeds in previously treated children with severe haemophilia A: results of the LEOPOLD Kids Trial. Haemophilia. 2016 May;22(3):354-60. doi: 10.1111/hae.12866. Epub 2015 Dec 9. PMID 26663410
- [Result] Keating GM. BAY 81-8973 (Octocog Alfa; Kovaltry(R)): A Review in Haemophilia A. BioDrugs. 2016 Oct;30(5):453-459. doi: 10.1007/s40259-016-0191-4. PMID 27577234
- [Result] Shah A, Delesen H, Garger S, Lalezari S. Pharmacokinetic properties of BAY 81-8973, a full-length recombinant factor VIII. Haemophilia. 2015 Nov;21(6):766-71. doi: 10.1111/hae.12691. Epub 2015 May 8. PMID 25952661
- [Result] Maas Enriquez M, Thrift J, Garger S, Katterle Y. BAY 81-8973, a full-length recombinant factor VIII: Human heat shock protein 70 improves the manufacturing process without affecting clinical safety. Protein Expr Purif. 2016 Nov;127:111-115. doi: 10.1016/j.pep.2016.07.009. Epub 2016 Jul 18. PMID 27436242
- [Result] Garmann D, McLeay S, Shah A, Vis P, Maas Enriquez M, Ploeger BA. Population pharmacokinetic characterization of BAY 81-8973, a full-length recombinant factor VIII: lessons learned - importance of including samples with factor VIII levels below the quantitation limit. Haemophilia. 2017 Jul;23(4):528-537. doi: 10.1111/hae.13192. Epub 2017 Feb 20. PMID 28220555
- [Result] Mahlangu JN, Ahuja SP, Windyga J, Church N, Shah A, Schwartz L. BAY 81-8973, a full-length recombinant factor VIII for the treatment of hemophilia A: product review. Ther Adv Hematol. 2018 Jul;9(7):191-205. doi: 10.1177/2040620718777903. Epub 2018 Jun 12. PMID 30013766
- [Result] Kenet G, Ljung R, Rusen L, Kerlin BA, Blanchette V, Saulyte Trakymiene S, Uscatescu V, Beckmann H, Tseneklidou-Stoeter D, Church N. Continued benefit demonstrated with BAY 81-8973 prophylaxis in previously treated children with severe haemophilia A: Interim analysis from the LEOPOLD Kids extension study. Thromb Res. 2020 May;189:96-101. doi: 10.1016/j.thromres.2020.03.005. Epub 2020 Mar 9. PMID 32197139
- [Result] Kenet G, Moulton T, Wicklund BM, Ahuja SP, Escobar M, Mahlangu J. Switching from Sucrose-Formulated rFVIII to Octocog Alfa (BAY 81-8973) Prophylaxis Improves Bleed Outcomes in the LEOPOLD Clinical Trials. J Blood Med. 2023 Jun 7;14:379-388. doi: 10.2147/JBM.S405624. eCollection 2023. PMID 37309365
- [Result] Ljung R, Chan AKC, Glosli H, Afonja O, Becker B, Tseneklidou-Stoeter D, Mancuso ME, Saulyte-Trakymiene S, Kenet G. BAY 81-8973 Efficacy and Safety in Previously Untreated and Minimally Treated Children with Severe Hemophilia A: The LEOPOLD Kids Trial. Thromb Haemost. 2023 Jan;123(1):27-39. doi: 10.1055/s-0042-1757876. Epub 2023 Jan 10. PMID 36626898
- [Derived] Ljung R, Chan AKC, Ahuja SP, Mancuso ME, Marquez JFC, Volk F, Blanchette V, Kerlin BA, Trakymiene SS, Glosli H, Kenet G. BAY 81-8973 Demonstrates Long-Term Safety and Efficacy in Children With Severe Haemophilia A: Results From the LEOPOLD Kids Extension Study. Eur J Haematol. 2025 Mar;114(3):556-565. doi: 10.1111/ejh.14362. Epub 2024 Dec 12. PMID 39667975
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 18 countries and consisted of: Part A - between 09-JUN-2011 (FPFV) and 02-JAN-2013 (LPLV); Part B - between 19-SEP-2012 (FPFV) and 09-SEP-2019 (LPLV); Extension study - between 21-DEC-2011 (FPFV) and 27-OCT-2020 (LPLV).
Pre-assignment Details: Overall, 58 participants were screened in Part A, of which 7 participants were screening failures and 51 participants received the study drug; 52 participants were screened in Part B, of which 9 participants were screening failures and 43 participants received the study drug. 46 participants from Part A and 36 from Part B entered the optional extension study.
Groups:
- PUPs/MTPs 0-<6 Years: Previously untreated patients (PUPs) or minimally treated patients (MTPs, patients who had no more than 3 exposure days [EDs] with any FVIII product) received BAY81-8973 15-50 IU/kg at least 1x/week for at least 50 EDs or until inhibitor development in main study - Part B. Participants having reached at least 50 EDs in main study - Part B were offered participation in an open label extension study and received BAY81-8973 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part B and extension study); participants who developed an inhibitor in main study - Part B were offered participation in open label extension study and received Immune Tolerance Induction (ITI) treatment with BAY81-8973 until successful eradication of the inhibitor, or until failure, for approximately 18 months.
Period: Main Study
Arm/Group | PTPs 0-12 Years | PUPs/MTPs 0-<6 Years
Started | 51 | 43
Started 0-<6 Years | 25 | 43
Started 6-12 Years | 26 | 0
Completed | 51 | 22
Not Completed | 0 | 21
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Inhibitor management | 0 | 17
Not completed — Withdrawal by Subject | 0 | 2
Period: Extension Study
Arm/Group | PTPs 0-12 Years | PUPs/MTPs 0-<6 Years
Started | 46 | 36
Completed | 45 | 25
Not Completed | 1 | 11
Not completed — Physician Decision | 0 | 1
Not completed — ITI therapy with marketed product | 0 | 1
Not completed — Incorrect visit planning | 0 | 1
Not completed — Family's decision | 0 | 1
Not completed — Failure of ITI therapy | 0 | 3
Not completed — Long travel | 0 | 1
Not completed — Diagnosed with von Willebrand disease | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Inhibitor management | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): all participants who entered Study Part A or Part B and received at least one infusion of study medication.
Groups:
- Main Study - Part A: PTPs 0-<6 Years: Previously treated patients (PTPs) aged below 6 years received BAY81-8973 25-50 IU/kg at least 2x/week for 6 months and at least 50 exposure days (ED) in main study - Part A.
- Main Study - Part A: PTPs 6-12 Years: Previously treated patients (PTPs) aged 6 to 12 years received BAY81-8973 25-50 IU/kg at least 2x/week for 6 months and at least 50 exposure days (ED) in main study - Part A.
- Main Study - Part B: PUPs/MTPs 0-<6 Years: Previously untreated patients (PUPs) or minimally treated patients (MTPs, patients who had no more then 3 exposure days (EDs) with any FVIII product) received BAY81-8973 15-50 IU/kg at least 1x/week for 50 EDs or until inhibitor development in main study - Part B.
- Total: Total of all reporting groups
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years | Total
Number analyzed (Participants) | 25 | 26 | 43 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.8 (1.3) | 8.8 (1.8) | 1.1 (0.8) | 3.9 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 25 | 26 | 43 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 9 | 10
  Not Hispanic or Latino | 23 | 25 | 34 | 82
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 24 | 37 | 85
  Black | 1 | 2 | 1 | 4
  American Indian or Alaska native | 0 | 0 | 1 | 1
  White, American Indian or Alaska native | 0 | 0 | 1 | 1
  Not reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of Total Bleeds Within 48 h
Description: Annualized number (mean +/- standard deviation) of total bleeds that occurred within 48 hours after all prophylaxis infusions (Part A: 6 months and at least 50 exposure days [EDs]; Part B: at least 50 EDs or until inhibitor development) was summarized and reported. Total bleeds: sum of spontaneous bleeds, trauma bleeds (only treated bleeds were classified as spontaneous or trauma), untreated bleeds and 'other' bleeds ('other' bleeds were infusions with reason given as 'other').
Time Frame: Within 48 hours post infusion
Population: Intent-to-treat (ITT) analysis set - main study: all participants of the SAF in main study who had infusion/bleeding data from the electronic patient diary (EPD)
Measure: Mean (Standard Deviation); unit: Bleeds
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 43
Bleeds | 2.23 (2.77) [lower limit 2.77] | 1.86 (3.08) [lower limit 3.08] | 1.9 (3.3) [lower limit 3.3]

2. Primary Outcome: Annualized Number of Total Bleeds Within 48 h
Description: Annualized number (median [inter-quartile range (Q1-Q3)]) of total bleeds that occurred within 48 hours after all prophylaxis infusions (Part A: 6 months and at least 50 exposure days [EDs]; Part B: at least 50 EDs or until inhibitor development) was summarized and reported. Total bleeds: sum of spontaneous bleeds, trauma bleeds (only treated bleeds were classified as spontaneous or trauma), untreated bleeds and 'other' bleeds ('other' bleeds were infusions with reason given as 'other').
Time Frame: Within 48 hours post infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Bleeds
Groups:
- Main Study - Part B: PUPs/MTPs 0-<6 Years: Previously untreated patients (PUPs) or minimally treated patients (MTPs, patients who had no more then 3 EDs with any FVIII product) received BAY81-8973 15-50 IU/kg at least 1x/week for 50 exposure days (ED) or until inhibitor development in main study - Part B.
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 43
Bleeds | 1.88 (0.00) [0.00 to 3.97] | 0.00 (0.00) [0.00 to 1.96] | 0.0 (0.0) [0.0 to 2.2]

3. Secondary Outcome: Annualized Number of Total Bleeds During Prophylaxis Treatment
Description: Annualized number (mean +/- standard deviation) of total bleeds that occurred during prophylaxis treatment was summarized and reported. Total bleeds: sum of spontaneous bleeds, trauma bleeds (only treated bleeds were classified as spontaneous or trauma), untreated bleeds and 'other' bleeds ('other' bleeds were infusions with reason given as 'other').
Time Frame: Part A: 6 months and at least 50 exposure days (EDs) (median 73 EDs; median 6 months); Part B: at least 50 EDs or until inhibitor development (median 46 EDs; median 8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bleeds
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 43
Bleeds | 4.16 (5.02) [lower limit 5.02] | 3.37 (5.01) [lower limit 5.01] | 7.1 (8.6) [lower limit 8.6]

4. Secondary Outcome: Annualized Number of Total Bleeds During Prophylaxis Treatment
Description: Annualized number (median [inter-quartile range (Q1-Q3)]) of total bleeds that occurred during prophylaxis treatment was summarized and reported. Total bleeds: sum of spontaneous bleeds, trauma bleeds (only treated bleeds were classified as spontaneous or trauma), untreated bleeds and 'other' bleeds ('other' bleeds were infusions with reason given as 'other').
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Bleeds
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 43
Bleeds | 2.03 (0.00) [0.00 to 6.02] | 0.93 (0.00) [0.00 to 5.77] | 4.7 (2.1) [2.1 to 8.9]

5. Secondary Outcome: Hemostatic Control During Major and Minor Surgeries
Description: For participants who underwent major or minor surgeries during the study, hemostasis during the surgeries was assessed as excellent, good, moderate or poor. Number of surgeries per assessment was summarized and reported.
Time Frame: as for outcome 3
Population: Participants in SAF in main study who underwent major or minor surgeries during the study
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 0 | 1 | 6
Number analyzed (Surgeries) | 0 | 1 | 6
Surgeries
  Minor surgery: number analyzed (Participants) | 0 | 0 | 5
  Minor surgery: number analyzed (Surgeries) | 0 | 0 | 5
  Minor surgery: Excellent | 0 | 0 | 3
  Minor surgery: Good | 0 | 0 | 1
  Minor surgery: Moderate | 0 | 0 | 0
  Minor surgery: Poor | 0 | 0 | 0
  Minor surgery: Not available | 0 | 0 | 1
  Major surgery: number analyzed (Participants) | 0 | 1 | 1
  Major surgery: number analyzed (Surgeries) | 0 | 1 | 1
  Major surgery: Excellent | 0 | 0 | 0
  Major surgery: Good | 0 | 1 | 1
  Major surgery: Moderate | 0 | 0 | 0
  Major surgery: Poor | 0 | 0 | 0
  Major surgery: Not available | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Inhibitor Development in Main Study
Description: Number of participants with confirmed positive FVIII inhibitor titer (≥ 0.6 Bethesda unit [BU/mL]) during the main study was summarized and classified as participants developing low titer inhibitor (i.e. ≥ 0.6 to ≤ 5.0 BU/mL) and participants developing high titer inhibitor (i.e. > 5.0 BU/mL).
Time Frame: as for outcome 3
Population: Participants in main study - safety analysis set (SAF, all participants who entered Study Part A or Part B and received at least one infusion of study medication) with inhibitor measurements done
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 42
Participants
  Low titer inhibitor | 0 | 0 | 6
  High titer inhibitor | 0 | 0 | 17

7. Secondary Outcome: Number of Participants With New Inhibitor Development in Extension Study
Description: Number of participants who had not developed an inhibitor during the main study but developed an inhibitor (confirmed positive FVIII inhibitor titer [≥ 0.6 BU/mL]) during the extension study was summarized and classified as participants developing low titer inhibitor (i.e. ≥ 0.6 to ≤ 5.0 BU/mL) and participants developing high titer inhibitor (i.e. > 5.0 BU/mL).
Time Frame: From start of extension study to at least 100 cumulative exposure days (EDs) (median 421 EDs; median 3.8 years)
Population: All participants who entered the extension study and had not developed inhibitors during the main study Part A or Part B
Measure: Count of Participants; unit: Participants
Groups:
- Extension Study - Former Part A Participants: Participants having reached at least 50 exposure days (EDs) in main study - Part A were offered participation in an open label extension study (optional). Participants who transitioned from main study - Part A to the extension study received BAY81-8973, 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part A and extension study).
- Extension Study - Former Part B Participants: Participants having reached at least 50 exposure days (EDs) in main study - Part B were offered participation in an open label extension study and received BAY81-8973 25-50 IU/kg at least 2x/week for at least 100 cumulative EDs (main study - Part B and extension study); participants who developed an inhibitor in main study - Part B were offered participation in open label extension study and received Immune Tolerance Induction (ITI) treatment with BAY81-8973 until successful eradication of the inhibitor, or until failure, for approximately 18 months.
Arm/Group | Extension Study - Former Part A Participants | Extension Study - Former Part B Participants
Number analyzed (Participants) | 46 | 16
Participants
  Low titer inhibitor (incl. false-positive) | 1 | 0
  High titer inhibitor | 0 | 0

8. Secondary Outcome: Factor VIII Recovery Values
Description: Incremental recovery of Factor VIII (FVIII) at 20-30 min after end of infusions was determined and mean recovery values were reported.
Time Frame: as for outcome 3
Population: Participants in intent-to-treat (ITT) analysis set in main study with valid FVIII recovery values
Measure: Mean (Standard Deviation); unit: International unit (IU)/dL per IU/kg
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 32
International unit (IU)/dL per IU/kg
  Participants without inhibitor: number analyzed (Participants) | 25 | 26 | 17
  Participants without inhibitor | 1.63 (0.31) | 1.72 (0.46) | 1.76 (0.55)
  Participants with low titer inhibitor: number analyzed (Participants) | 0 | 0 | 4
  Participants with low titer inhibitor |  |  | 0.86 (0.56)
  Participants with high titer inhibitor: number analyzed (Participants) | 0 | 0 | 11
  Participants with high titer inhibitor |  |  | 0.38 (0.42)

9. Secondary Outcome: Consumption of Factor VIII in All Infusions
Description: Factor VIII (FVIII) usage/consumption was summarized for all infusions. Consumption per participant's body weight per year was calculated and reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: international units/kilogram/year
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 43
international units/kilogram/year | 5499.1 (1996.2) [lower limit 1996.2] | 4679.1 (1688.7) [lower limit 1688.7] | 2195.8 (1903.6) [lower limit 1903.6]

10. Secondary Outcome: Consumption of FVIII in Infusions for Prophylaxis
Description: Factor VIII (FVIII) usage/consumption was summarized for prophylaxis infusions. Consumption per participant's body weight per year was calculated and reported.
Time Frame: as for outcome 3
Population: Participants in intent-to-treat (ITT) analysis set in main study with at least one dose of prophylaxis treatment with study drug
Measure: Mean (Standard Deviation); unit: international units/kilogram/year
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 25 | 26 | 42
international units/kilogram/year | 5224.8 (1760.2) [lower limit 1760.2] | 4492.7 (1667.6) [lower limit 1667.6] | 1486.6 (963.3) [lower limit 963.3]

11. Secondary Outcome: Consumption of FVIII in Infusions for the Treatment of Bleeds
Description: Factor VIII (FVIII) usage/consumption was summarized for infusions used to treat breakthrough bleeds. Consumption per participant's body weight per year was calculated and reported.
Time Frame: as for outcome 3
Population: Participants in intent-to-treat (ITT) analysis set in main study with at least one bleed treated with study drug
Measure: Mean (Standard Deviation); unit: international units/kilogram/year
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 15 | 11 | 35
international units/kilogram/year | 457.07 (526.87) [lower limit 526.87] | 391.64 (219.61) [lower limit 219.61] | 835.4 (1926.4) [lower limit 1926.4]

12. Secondary Outcome: Number of Infusions Per Bleed
Description: The number of infusions used to treat a bleed was defined as the first infusion to treat the bleed plus all follow-up infusions to treat the same bleed, if any. The mean value of number of infusions for each bleed was calculated and reported.
Time Frame: as for outcome 3
Population: Participants in intent-to-treat (ITT) analysis set in main study with at least one bleed
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 15 | 13 | 37
Infusions | 1.3 (1.8) [lower limit 1.8] | 1.4 (1.7) [lower limit 1.7] | 1.7 (8.7) [lower limit 8.7]

13. Secondary Outcome: Response to Treatment of Bleeds
Description: Participants or caregivers were asked to assess the response to treatment of bleeds as excellent, good, moderate or poor. Percentage of bleeds per assessment was summarized and reported.
Time Frame: as for outcome 3
Population: Participants in intent-to-treat (ITT) analysis set in main study with at least one bleed
Measure: Count of Units; unit: Bleeds assessed for the response
Units Other Than Participants: Bleeds assessed for the response
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years
Number analyzed (Participants) | 15 | 13 | 37
Number analyzed (Bleeds assessed for the response) | 44 | 37 | 105
Bleeds assessed for the response
  Excellent | 20 | 12 | 27
  Good | 23 | 18 | 56
  Moderate | 0 | 7 | 16
  Poor | 1 | 0 | 6

14. Secondary Outcome: Half-life (t1/2) of BAY81-8973 in Plasma
Description: Half-life (t1/2) of BAY81-8973 in plasma was measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Pre-infusion and until 24 hours post infusion
Population: Participants in PK analysis set (PKS) - A with evaluable data for this endpoint (PKS - A: all participants who entered main study - Part A and received at least one infusion of study medication with evaluable pharmacokinetic data)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years
Number analyzed (Participants) | 2 | 9
Hours | 13.2 (39.7) | 12.1 (16.3)

ADVERSE EVENTS:
Time Frame: Main study - Part A: from the first BAY81-8973 infusion until 3 days after the last infusion (median 6 months); Main study - Part B: from the first BAY81-8973 infusion until 7 days after the last infusion (median 8 months); Extension: from start of extension study until 3 days after the last infusion in extension study (median 3.1 years)
Arm/Group | Main Study - Part A: PTPs 0-<6 Years | Main Study - Part A: PTPs 6-12 Years | Main Study - Part B: PUPs/MTPs 0-<6 Years | Extension Study - Former Part A Participants | Extension Study - Former Part B Participants
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/43 | 0/46 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/25 | 5/26 | 26/43 | 23/46 | 14/36
Other Adverse Events (participants affected / at risk) | 16/25 | 19/26 | 28/43 | 41/46 | 24/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Part A: PTPs 0-<6 Years (N=25) | Main Study - Part A: PTPs 6-12 Years (N=26) | Main Study - Part B: PUPs/MTPs 0-<6 Years (N=43) | Extension Study - Former Part A Participants (N=46) | Extension Study - Former Part B Participants (N=36)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Factor VIII inhibition (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epidemic pleurodynia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anti factor VIII antibody positive (Investigations) | 0 (0) | 0 (0) | 22 (24) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electroencephalogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 3 (3)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Internal device exposed (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenotonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Dental cleaning (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune tolerance induction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Part A: PTPs 0-<6 Years (N=25) | Main Study - Part A: PTPs 6-12 Years (N=26) | Main Study - Part B: PUPs/MTPs 0-<6 Years (N=43) | Extension Study - Former Part A Participants (N=46) | Extension Study - Former Part B Participants (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 3 (10)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 2 (2)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (2) | 6 (8) | 5 (5) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (8) | 4 (4) | 6 (10)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 5 (10) | 2 (2) | 12 (19) | 8 (19) | 11 (21)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 3 (5)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 2 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (4)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hookworm infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (2) | 6 (16) | 13 (31) | 9 (23)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (3)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (10) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 6 (8) | 1 (3)
Tonsillitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 10 (25) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3) | 6 (11) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Viral infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 6 (15) | 2 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Genital contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 9 (11) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (9) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 0 (0) | 8 (23) | 0 (0)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (4) | 1 (1) | 9 (18) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 5 (8) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 3 (3) | 3 (3) | 1 (3)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (3) | 0 (0) | 2 (5) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the small number of participants per reporting group, all presented summary measures (e.g. mean and proportion) have to be evaluated with caution. If displayed standard deviation should be taken into account. The participant who had a low titer inhibitor detected after 549 EDs during the extension study was considered to have a false positive result due to cross reactivity with IgG anticardiolipin antibodies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results within 60 days. The sponsor can require changes to the communication for any patentable subject matter or termed confidential information. The PI cannot publish the results prior the first multicenter publication. If there is no multicenter publication within 18 months after the trial completion the PI has the right to publish the results from the PI site

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT01311648/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT01311648/SAP_001.pdf